CLINICAL TRIAL: NCT06826742
Title: Intravenous Methadone Versus Intrathecal Morphine for Analgesia Following Cesarean Delivery: a Randomized Clinical Trial
Brief Title: Intravenous Methadone Versus Intrathecal Morphine for Analgesia Following Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Emily E. Sharpe, M.D., Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-000215
Record Dates: First submitted 2025-02-10; First posted 2025-02-14 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Cesarean Delivery
Keywords: methadone; morphine; intrathecal; cesarean
MeSH Terms: interventions — Methadone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Spinal Anesthesia with Intravenous Methadone (Experimental): Subjects will receive spinal anesthesia (intrathecal bupivacaine with fentanyl) with intravenous methadone
  Interventions: Drug: Intravenous line (IV) Methadone
- Spinal Anesthesia with Intrathecal Morphine (Active Comparator): Subjects will receive spinal anesthesia (intrathecal bupivacaine with fentanyl) with intrathecal morphine
  Interventions: Drug: Intrathecal Morphine

INTERVENTIONS:
Drug: Intravenous line (IV) Methadone — Subjects will receive standardized spinal anesthesia without intrathecal morphine (intrathecal 1.6-2 mL 0.75% bupivacaine + dextrose, 15 mcg fentanyl) and intravenous methadone (0.2mg/kg total body weight up to max dose of 20 mg, with saline added to make total volume 2 mL)
  The Intravenous line (IV) methadone will be administered after cord clamping and administration of uterotonics with the dose of medication divided into 4 equal aliquots each administered 5 minutes apart.
  Arms: Spinal Anesthesia with Intravenous Methadone
Drug: Intrathecal Morphine — Subjects will receive standardized spinal anesthesia with intrathecal morphine 150 micrograms and no methadone (2cc dose of IV normal saline)
  The Intravenous line (IV) saline will be administered after cord clamping and administration of uterotonics with the dose of medication divided into 4 equal aliquots each administered 5 minutes apart.
  Arms: Spinal Anesthesia with Intrathecal Morphine

SUMMARY:
The purpose of this study is to determine if there is a difference in opioid requirements at 0-48 hours after scheduled cesarean delivery in patients receiving 150 mcg intrathecal morphine compared to 0.2 mg/kg (maximum 20 mg) intravenous methadone.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age over 18 years old
* Scheduled cesarean delivery

Exclusion Criteria:

* Any contraindication to the administration of a spinal technique for anesthesia
* History of intolerance or adverse reaction to opioid medications
* History of chronic pain, opioid use >30 OME/day, or substance use disorder
* History of obstructive sleep apnea, chronic obstructive pulmonary disease, or respiratory compromise (SpO2 <92% on room air, or has a pre-existing oxygen requirement)
* History of liver or kidney failure
* Diagnosis of pre-eclampsia with current pregnancy
* Depression requiring more than one medication
* Planned use of CSE technique
* BMI >50.0 kg/m2
* ASA status IV, V
* No prior history of an ECG demonstrating QTc > 440ms
* Surgical complication requiring conversion to general anesthesia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-02-12 (Actual); Primary Completion 2025-09-14 (Actual); Study Completion 2025-09-23 (Actual)

PRIMARY OUTCOMES:
Total opioid consumption | 24 hours post-delivery, 48 hours post-delivery
  Total opioid consumption of either intrathecal opiate or intravenous methadone at 24-48 hours after delivery.

SECONDARY OUTCOMES:
Obstetric Quality of Recovery-10 (ObsQoR-10) Scoring Tool | 24 hours, 48 hours, 7 days
  The Obstetric Quality of Recovery-10 (ObsQoR-10), is a patient-reported 10-item questionnaire used to assess quality of recovery following spinal administration of pain medication. Patients rate each recovery item on a scale of 0 to 10, with 0 = worst possible recovery and 10 = best possible recovery. Total score ranges from 0-100 with higher scores indicating a better recovery after childbirth.
Numeric Rating Scale (NRS) pain score at rest | 12 hours, 24 hours, 36 hours, 48 hours, 7 days
  A Numeric Rating Scale (NRS) for pain is a patient-reported item regarding the level of pain experienced at rest and is measured on a Likert scale from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable".
Numeric Rating Scale (NRS) for movement-evoked pain | 12 hours, 24 hours, 36 hours, 48 hours, 7 days
  A Numeric Rating Scale (NRS) score for movement-evoked pain is a patient-reported item regarding the level of pain experienced with provoking maneuvers such as cough, inspiration/expiration, sitting up, knee flexion, hip flexion, rolling over in bed, and walking. The NRS is measured on a Likert scale from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable".
Numeric Rating Scale (NRS) for pain in previous 24 hours | 12 hours, 24 hours, 36 hours, 48 hours, 7 days
  A Numeric Rating Scale (NRS) score for highest level of pain is a patient-reported item regarding the level of pain experienced in the last 24 hours. The NRS is measured on a Likert scale from 0 to 10, where 0 represents "no pain" and 10 represents "the worst pain imaginable".
Pruritus | 12 hours, 24 hours, 36 hours, 48 hours
  The severity of pruritus post spinal administration will be patient-reported on a 4-point Likert scale where 0 = none and 3 = severe.
Richmond Agitation Sedation Scale (RASS) | 12 hours, 24 hours, 36 hours, 48 hours
  The Richmond Agitation Sedation Scale (RASS) will be used to assess the level of alertness and agitated behavior in patients. The patient's level of consciousness and sedation are rated by care provider, ranging from a combative state (+4) to an unarousable state (-5), with a "calm and alert" score at 0.

CONTACTS AND LOCATIONS:
Overall Officials: Emily E Sharpe, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials